CLINICAL TRIAL: NCT04076111
Title: Patterns of Breast Cancer Management and Prognosis of Breast Cancer in China：a Multicenter, Prospective, Real-world Cohort Study
Brief Title: Patterns of Breast Cancer Management and Prognosis of Breast Cancer in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fengxi Su (Other)
Responsible Party: Sponsor-Investigator, Fengxi Su, PI, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Other Study IDs: BCSCO003
Record Dates: First submitted 2019-08-25; First posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter, prospective, e, real-world cohort survey initiated by researchers to focus on the patterns of breast cancer management and prognosis of breast cancer in China, and to establish the multicenter, prospective breast cancer data platform. A total of 18 sites in Guangdong and Henan have cooperated to build a cooperative network unit. The sites will conduct prospective and standardized records concerning the clinical pathological features, treatment and prognosis of the early breast cancer patients who are treated in their own site each year, registering in the REDCap system.This real-world cohort study aims to provide a representative and reliable survey data of epidemiological characteristics, clinical treatment and prognosis of patients with early breast cancer in China and explore the establishment of a national multi-center breast cancer data platform model.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are hospitalized and treated in a collaborative network unit
* Agree to enroll in the study and sign the informed consent form
* Histological diagnosis of ductal carcinoma in situ or invasive breast cancer
* Accept the Surgery-based surgical treatment
* Willing to cooperate with follow-up work

Exclusion Criteria:

* Previously Excisional biopsy (including minimally invasive resection) of the patient's breast
* Previously received neoadjuvant chemotherapy
* Imaging or histological evidence of distant metastasis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had early stage breast cancer and completed breast surgery
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2019-09-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Breast-conserving surgery rate, | baseline
  the proportion between breast-conserving surgery and breast mastectomy surgery baseline
Breast-conserving surgery rate, sentinel lymph node biopsy rate | baseline
  the proportion between sentinel lymph node biopsy and axillary lymph node dissection

SECONDARY OUTCOMES:
Epidemiological distribution of pathological stage of breast cancer | baseline
  the American Joint Committee on Cancer(AJCC) cancer staging system is used to assign stage for breast cancer patients,including primary tumor stage, regional nodes stage and metastasis stage
Disease free survival (DFS) | 5year
  Disease free survival (DFS), which defined as the time from the diagnosis of breast cancer to the confirmed time of metastatic disease, or death due to any other cause.
Overall survival (OS) | 5year
  Overall survival (OS), which defined as the time from the beginning of diagnosis of breast cancer to the death with any causes.

CONTACTS AND LOCATIONS:
Overall Officials: Fengxi Su, MD, Study Chair — Sun Yat-sen Menorial Hospital; Qiang liu, MD, Study Chair — Sun Yat-sen Menorial Hospital; Musheng Zeng, MD, Study Director — Sun Yat-sen University; Qianjun Chen, MD, Study Director — Guuangdong Province Hospital of Chinese Medicine
Locations (5):
- China (5):
  - Guangdong Province Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital,Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Cancer Hospital OF Shantou University Medical College, Shantou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan